CLINICAL TRIAL: NCT05428839
Title: The PREDICTOR Study: Assessing Diagnostic Predictors of Airway Collapse in Patients With Obstructive Sleep Apnea
Acronym: PREDICTOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20021-003
Record Dates: First submitted 2022-05-10; First posted 2022-06-23 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-03

CONDITIONS: Sleep Apnea, Obstructive
Keywords: OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Pharyngeal width measurement — A simple, non-invasive measurement of the pharyngeal width inside each subjects mouth

SUMMARY:
This study is an exploratory, multicenter study of up to 300 subjects diagnosed with obstructive sleep apnea who are being evaluated for airway surgery. Subjects will undergo standard evaluation for airway surgery as part of standard of care. In addition to the standard airway assessment, a simple, non-invasive measurement of the width of the inside of each subjects mouth will be performed. This measurement takes 2-3 minutes to perform.

DETAILED DESCRIPTION:
The objective of the study is to determine whether pharyngeal width (inside of the mouth) is an appropriate measurement to predict absence of complete concentric collapse (CCC) at the soft palate

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the indications for the Inspire Upper Airway Stimulation
* Patient is being evaluated by drug-induced sleep endoscopy as standard-of-care diagnostic for OSA surgery.

Exclusion Criteria:

* Patient is unable to lie supine for 2-3 minutes in order to undergo airway measurement
* Any other reason the investigator deems that the patient is unfit for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of pharyngeal width to determine if there is correlation between pharyngeal width and presence or absence of complete concentric collapse at the soft palate during drug induced sleep endoscopy | Baseline, prior to routine diagnostic drug induced sleep endoscopy
  Pharyngeal width will be measured in millimeters using a caliper

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Valley ENT, Scottsdale, Arizona
  - Rush University Medical Center, Chicago, Illinois
  - Mason City Clinic, Mason City, Iowa
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - ENT Specialty Care of MN, Saint Louis Park, Minnesota
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No